CLINICAL TRIAL: NCT06470451
Title: A Confirmatory Phase 3 Multicenter, Randomized, Double-Blind, Placebo-Controlled Study of the Efficacy of Topical HyBryte™ (Hypericin Sodium) and Visible-Light Activation for the Treatment of Cutaneous T-Cell Lymphoma (CTCL)
Brief Title: Confirmatory Study of Topical HyBryte™ vs. Placebo for the Treatment of CTCL
Acronym: FLASH2
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Soligenix (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HPN-CTCL-03-EUR
Record Dates: First submitted 2024-06-17; First posted 2024-06-24 (Actual); Last update posted 2025-11-14 (Actual); Status verified 2025-11

CONDITIONS: CTCL/ Mycosis Fungoides; CTCL; Mycosis Fungoides; Cutaneous T Cell Lymphoma
MeSH Terms: conditions — Mycosis Fungoides; Lymphoma, T-Cell, Cutaneous | interventions — hypericin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- HyBryte (0.25% Hypericin) (Experimental): HyBryte gel is applied twice weekly for 18 weeks.
  Interventions: Drug: Hypericin
- Placebo (Placebo Comparator): Placebo gel is indistinguishable from HyBryte gel, and is applied twice weekly for 18 weeks.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Hypericin — HyBryte gel (0.25% hypericin) is applied twice weekly for 18 weeks. Treated lesions are covered with opaque material (such as opaque clothing), followed 21 (±3) hours later by the administration of visible light.
  Other Names: HyBryte; SGX301
  Arms: HyBryte (0.25% Hypericin)
Drug: Placebo — Placebo gel is applied twice weekly for 18 weeks. Treated lesions are covered with opaque material (such as opaque clothing), followed 21 (±3) hours later by the administration of visible light.
  Arms: Placebo

SUMMARY:
To evaluate the use of HyBryte, a topical photosensitizing agent, to treat patients with patch/plaque phase cutaneous T-cell lymphoma (mycosis fungoides).

DETAILED DESCRIPTION:
The primary objective of this Phase 3 study is to evaluate the ability of an 18-week course of HyBryte and visible light to induce a Treatment Response in patients with patch/plaque phase CTCL compared to patients receiving placebo and visible light.The study will evaluate the efficacy and safety of HyBryte (0.25% hypericin) gel or placebo gel applied twice weekly for 18 weeks. Treated lesions will be covered with opaque material (such as opaque clothing), followed 21 (±3) hours later by the administration of visible light. All of the participant's lesions that are readily available for exposure to the visible light source will be treated and 3 to 5 index lesions in each patient will be prospectively identified and documented for modified Composite Assessment of Index Lesion Severity (mCAILS) evaluation. Participants will be followed every 4 weeks for a total of 12 weeks following their last light session.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have a clinical diagnosis of cutaneous T-cell lymphoma (CTCL), Stage IA, Stage IB, or Stage IIA.
* Patients with a minimum of three (3) evaluable, discrete lesions.
* Patients willing to follow the clinical protocol and voluntarily give their written informed consent.
* Female patients not pregnant or nursing and willing to undergo a pregnancy test within 30 days prior to treatment initiation.

Exclusion Criteria:

* History of sun hypersensitivity and photosensitive dermatoses including porphyria, systemic lupus erythematosus, Sjögren's syndrome, xeroderma pigmentosum, polymorphous light eruptions, or radiation therapy within 30 days of enrolling.
* History of allergy or hypersensitivity to any of the components of HyBryte.
* A Screening ECG with a QT interval >470 ms (corrected for heart rate using the Fridericia's formula).
* All women of childbearing potential (WOCBP) and males with female partners who are WOCBP not willing to use effective contraception.
* Patients receiving topical steroids or other topical treatments (eg, nitrogen mustard) on treated lesions for CTCL within 2 weeks of enrollment.
* Patients receiving systemic steroids, psoralen UVA radiation therapy (PUVA), narrow band UVB light therapy (NB-UVB) or carmustine (BCNU) or other systemic therapies for CTCL within 4 weeks of enrollment.
* Patients who have received electron beam irradiation within 3 months of enrollment.
* Patients with a history of significant systemic immunosuppression.
* Patients taking other investigational drugs or drugs of abuse within 30 days of entry into this study.
* Patients whose condition is spontaneously improving.
* Patients with tumor stage or erythrodermic CTCL (stages IIB-IV).
* Patients with extensive skin disease (>30% body surface area) who would be, in the judgement of the Principal Investigator, candidates for systemic treatment.
* Patient has any condition that, in the judgment of the PI, is likely to interfere with participation in the study.
* Prior participation in the current study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2025-01-07 (Actual); Primary Completion 2026-07 (Estimated); Study Completion 2026-10 (Estimated)

PRIMARY OUTCOMES:
Number of Participants with a Treatment Response in the Modified Composite Assessment of Index Lesion Disease Severity (mCAILS) score | 18 weeks
  A treatment response is defined as a ≥50% improvement in the cumulative mCAILS score of the index lesions at Week 18 when compared to the mCAILS score at baseline.
  The Modified Composite Assessment of Index Lesion Disease Severity (mCAILS) score measures: Erythema (or redness) on a scale of 0 (no redness) to 8 (very red), Scaling on a scale of 0 (no scaling) to 8 (all of the lesion is covered by a very rough surface), Plaque Elevation on a scale of 0 (no evidence of plaque above normal skin level) to 3 (plaque shows marked elevation above normal skin level) and Surface Area on a scale of 0 (no lesion/surface area is 0 cm^2) to 18 (the lesion is larger than 300 cm^2). A lower score means a better outcome.

SECONDARY OUTCOMES:
Patch Lesion Response Rates | 18 weeks
  The proportion of patch lesions achieving a treatment response at Week 18. A treatment response is defined as a ≥50% improvement in mCAILS score when compared to the mCAILS score at baseline for individual lesions.
  The Modified Composite Assessment of Index Lesion Disease Severity (mCAILS) score is measured as previously described.
Plaque Lesion Response Rates | 18 weeks
  The proportion of plaque lesions achieving a treatment response at Week 18. A treatment response is defined as a ≥50% improvement in mCAILS score when compared to the mCAILS score at baseline for individual lesions.
  The Modified Composite Assessment of Index Lesion Disease Severity (mCAILS) score is measured as previously described.

CONTACTS AND LOCATIONS:
Locations (17):
- United States (17):
  - Medical Dermatology Specialists, Phoenix, Arizona
  - Mayo Clinic, Scottsdale, Arizona
  - Therapeutics Clinical Research, San Diego, California
  - University of South Florida, Tampa, Florida
  - Northwestern University, Chicago, Illinois
  - Dawes Fretzin Dermatology Group, Indianapolis, Indiana
  - Washington University, St Louis, Missouri
  - Rochester Skin Lymphoma Medical Group, Fairport, New York
  - Columbia University Medical Center, New York, New York
  - Accellacare (PMG), Wilmington, North Carolina
  - Penn State Health Hershey Medical Center, Hershey, Pennsylvania
  - Hospital of the University of Pennsylvania, Philadelphia, Pennsylvania
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania
  - Vanderbilt University, Nashville, Tennessee
  - MD Anderson, Houston, Texas
  - Austin Institute for Clinical Research, Pflugerville, Texas
  - Inova Schar Cancer Institute, Fairfax, Virginia

IPD SHARING:
Plan to Share IPD: No